CLINICAL TRIAL: NCT01458015
Title: Phase 4 Study of Tapentadol vs Oxycodone in Neuropathic Pain
Brief Title: Tapentadol Versus Oxycodone - a Mechanism-based Treatment Approach in Neuropathic Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Ralf Baron, Prof. Dr. med., University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TapOxy01
Record Dates: First submitted 2011-08-05; First posted 2011-10-24 (Estimated); Results first posted 2024-12-17 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Neuropathy
Keywords: QST (quantitative sensory testing); neuropathic pain; tapentadol pr; oxycodone
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neuralgia | interventions — Tapentadol; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxycodone (Active Comparator)
  Interventions: Drug: tapentadol, oxycodone
- tapentadol (Active Comparator)
  Interventions: Drug: tapentadol, oxycodone

INTERVENTIONS:
Drug: tapentadol, oxycodone — tapentadol pr 100-500 mg oxycodone cr 20-120mg
  Other Names: Palexia

SUMMARY:
The purpose of this study is to elucidate whether the additional mechanism of analgesia, i.e. reuptake inhibition of norepinephrine, of tapentadol leads to a change in different pain signs and symptoms in comparison to oxycodone.

ELIGIBILITY:
Inclusion Criteria:

* thermal or mechanical hyperalgesia
* chronic neuropathic pain (NRS => 6)

Exclusion Criteria:

* non-specific

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Baron, Prof. Dr., Principal Investigator — Head of Unit of Neuropathic Pain Research and Therapy, Department of Neurology, University Clinic Kiel
Locations (1):
- Division for Neurological Pain Research and Therapy, Kiel, Schleswig-Holstein, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Tapentadol: received 200-500 mg Tapentadol PR (prolonged release), individual titration
- Oxycodon Retard: received 40-120 mg Oxycodon CR (controled release), individual titration
Period: Overall Study
Arm/Group | Tapentadol | Oxycodon Retard
Started | 2 | 1
Completed | 2 | 0
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxycodone | Tapentadol | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 57 [57 to 57] | 52 [47 to 57] | 53.6 [47 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  caucasian/european | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Germany | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Pain Threshold (MPT)
Description: Change of Mechanical Pain Threshold from baseline to V6 The mechanical pain threshold (MPT) was measured according to the established protocol of Deutscher Forschungsverbund Neuropathischer Schmerz (DFNS). See Rolke, R et al. "Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values." Pain vol. 123,3 (2006): 231.
  Logarithmically transformed raw data were z-transformed by subtracting the mean value of the corresponding reference group followed by a division the respective standard deviation. If the resulting z-value exceeds 1.96, it is outside the 95% confidence interval of the standard normal distribution with zero mean and unit variance, independent of the original units of measurement.
  (also see Rolke et. al.) A lower z-value indicates an improvement.
Time Frame: day 0 (baseline) and day 78 (V6; 10 weeks)
Population: Due to low number of participants only descriptive data is available
Measure: Mean (Full Range); unit: Z-score
Arm/Group | Oxycodone | Tapentadol
Number analyzed (Participants) | 1 | 2
Z-score
  V1 | 1.1 [1.1 to 1.1] | 2.6 [2.2 to 3]
  V6: number analyzed (Participants) | 0 | 2
  V6 |  | 0.55 [-1.9 to 3]

2. Primary Outcome: Heat Pain Threshold (HPT)
Description: Change of Heat Pain Threshold from V1 to V6 The was Heat Pain Threshold (HPT)measured according to the established protocol of Deutscher Forschungsverbund Neuropathischer Schmerz (DFNS). See Rolke, R et al. "Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values." Pain vol. 123,3 (2006): 231.
  Raw data were z-transformed by subtracting the mean value of the corresponding reference group followed by a division the respective standard deviation. If the resulting z-value exceeds 1.96, it is outside the 95% confidence interval of the standard normal distribution with zero mean and unit variance, independent of the original units of measurement.
  (also see Rolke et. al.) A lower z-value indicates an improvement.
Time Frame: day 0 (baseline) and day 78 (10 weeks)
Population: Due to low number of participants only descriptive data is available
Measure: Mean (Full Range); unit: Z-score
Groups:
- Tapentadol: received 200-500 mg Tapentadol PR, individual titration
- Oxycodone: received 40-120 mg Oxycodone CR, individual titration
Arm/Group | Tapentadol | Oxycodone
Number analyzed (Participants) | 2 | 1
Z-score
  V1 | -0.5 [-1.8 to 2.8] | -0.2 [-0.2 to -0.2]
  V6: number analyzed (Participants) | 2 | 0
  V6 | -1.4 [-1.9 to -0.9] |

3. Primary Outcome: Wind-Up Ratio (WUR)
Description: Change of Wind-Up Ratio from V1 to V6 The Wind-Up Ratio (WUR) was measured according to the established protocol of Deutscher Forschungsverbund Neuropathischer Schmerz (DFNS). See Rolke, R et al. "Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values." Pain vol. 123,3 (2006): 231.
  Logarithmically transformed raw data were z-transformed by subtracting the mean value of the corresponding reference group followed by a division the respective standard deviation. If the resulting z-value exceeds 1.96, it is outside the 95% confidence interval of the standard normal distribution with zero mean and unit variance, independent of the original units of measurement.
  (also see Rolke et. al.) A lower z-value indicates an improvement.
Time Frame: day 0 (baseline) and day 78 (10 weeks)
Population: Due to low number of participants only descriptive data is available
Measure: Mean (Full Range); unit: Z-score
Arm/Group | Tapentadol | Oxycodone
Number analyzed (Participants) | 2 | 1
Z-score
  V1 | -0.6 [-0.8 to -0.4] | -0.2 [-0.2 to -0.2]
  V6: number analyzed (Participants) | 2 | 0
  V6 | 0.75 [-0.6 to 2.1] |

4. Primary Outcome: Cold Pain Threshold (CPT)
Description: Change of Cold Pain Threshold from baseline to V6 The Cold Pain Threshold (CPT) was measured according to the established protocol of Deutscher Forschungsverbund Neuropathischer Schmerz (DFNS). See Rolke, R et al. "Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values." Pain vol. 123,3 (2006): 231.
  Raw data were z-transformed by subtracting the mean value of the corresponding reference group followed by a division the respective standard deviation. If the resulting z-value exceeds 1.96, it is outside the 95% confidence interval of the standard normal distribution with zero mean and unit variance, independent of the original units of measurement.
  (also see Rolke et. al.) A lower z-value indicates an improvement.
Time Frame: day 0 (baseline) and day 78 (10 weeks)
Population: Due to low recruitement numbers only descriptive data is available
Measure: Mean (Full Range); unit: Z-score
Arm/Group | Tapentadol | Oxycodone
Number analyzed (Participants) | 2 | 1
Z-score
  V1 | 0.35 [-1.2 to 1.9] | -1.1 [-1.1 to -1.1]
  V6: number analyzed (Participants) | 2 | 0
  V6 | 0.35 [-1.2 to 1.9] |

5. Primary Outcome: Pressure Pain Threshold (PPT)
Description: Change of Pressure Pain Threshold from V1 to V6 The Pressure Pain Threshold (PPT) was measured according to the established protocol of Deutscher Forschungsverbund Neuropathischer Schmerz (DFNS). See Rolke, R et al. "Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values." Pain vol. 123,3 (2006): 231.
  Logarithmically transformed raw data were z-transformed by subtracting the mean value of the corresponding reference group followed by a division the respective standard deviation. If the resulting z-value exceeds 1.96, it is outside the 95% confidence interval of the standard normal distribution with zero mean and unit variance, independent of the original units of measurement.
  (also see Rolke et. al.) A lower z-value indicates an improvement.
Time Frame: day 0 (baseline) and day 78 (V6; 10 weeks)
Population: Due to low number of participants only descriptive data is available
Measure: Mean (Full Range); unit: Z-score
Arm/Group | Oxycodone | Tapentadol
Number analyzed (Participants) | 1 | 2
Z-score
  V1 | 0 [0 to 0] | 1.65 [-1.9 to 5.2]
  V6: number analyzed (Participants) | 0 | 2
  V6 |  | 0.9 [-3.1 to 4.9]

6. Primary Outcome: Mechanical Pain Sensitivity (MPS)
Description: Change of Mechanical Pain Sensitivity from V1 to V6 The Mechanical Pain Sensitivity (MPS) was measured according to the established protocol of Deutscher Forschungsverbund Neuropathischer Schmerz (DFNS). See Rolke, R et al. "Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values." Pain vol. 123,3 (2006): 231.
  Logarithmically transformed raw data were z-transformed by subtracting the mean value of the corresponding reference group followed by a division the respective standard deviation. If the resulting z-value exceeds 1.96, it is outside the 95% confidence interval of the standard normal distribution with zero mean and unit variance, independent of the original units of measurement.
  (also see Rolke et. al.) A lower z-value indicates an improvement.
Time Frame: day 0 (baseline) and day 78 (V6; 10 weeks)
Population: Due to low number of participants only descriptive data is available
Measure: Mean (Full Range); unit: Z-score
Arm/Group | Oxycodone | Tapentadol
Number analyzed (Participants) | 1 | 2
Z-score
  V1 | 2.2 [2.2 to 2.2] | 2 [1.8 to 2.2]
  V6 | -0.4 [-0.4 to -0.4] | 1.5 [-0.9 to 3.9]

7. Primary Outcome: Dynamic Mechanical Allodynia (DMA)
Description: Change of Dynamic Mechanical Allodynia from V1 to V6 The Dynamic Mechanical Allodynia (DMA) was measured according to the established protocol of Deutscher Forschungsverbund Neuropathischer Schmerz (DFNS). "Subjects were asked to give a pain rating for each stimulus on a '0-100' numerical rating scale ('0' indicating "no pain", and '100' indicating "most intense pain imaginable")." See Rolke, R et al. "Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values." Pain vol. 123,3 (2006): 231.
  A lower score indicates an improvement.
Time Frame: day 0 (baseline) and day 78 (V6; 10 weeks)
Population: Due to low number of participants only descriptive data is available
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Oxycodone | Tapentadol
Number analyzed (Participants) | 1 | 2
score on a scale
  V1 | 41 [41 to 41] | 44 [40 to 48]
  V6 | 2 [2 to 2] | 5 [1 to 9]

8. Primary Outcome: Pain Upon Numeric Rating Scale
Description: Change of pain upon Numeric Rating Scale (NRS; 0 = no pain at all; 10 = maximum pain imaginable) from V1 to V6
Time Frame: day 0 (baseline) and day 78 (V6; 10 weeks)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Oxycodone | Tapentadol
Number analyzed (Participants) | 1 | 2
score on a scale
  V1 | 6 [6 to 6] | 9.5 [9 to 10]
  V6 | 3 [3 to 3] | 5.5 [4 to 7]

9. Secondary Outcome: Cold Detection Threshold (CDT)
Description: Change of Cold Detection Threshold from V1 to V6 The Cold Detection Threshold (CDT) was measured according to the established protocol of Deutscher Forschungsverbund Neuropathischer Schmerz (DFNS). See Rolke, R et al. "Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values." Pain vol. 123,3 (2006): 231.
  Raw data were z-transformed by subtracting the mean value of the corresponding reference group followed by a division the respective standard deviation. If the resulting z-value exceeds 1.96, it is outside the 95% confidence interval of the standard normal distribution with zero mean and unit variance, independent of the original units of measurement.
  (also see Rolke et. al.). A higher z-value indicates an improvement.
Time Frame: day 0 (baseline) and day 78 (10 weeks)
Population: Due to low number of participants only descriptive data can be provided.
Measure: Mean (Full Range); unit: Z-score
Arm/Group | Tapentadol | Oxycodone
Number analyzed (Participants) | 2 | 1
Z-score
  V1 | -1.2 [-2 to -0.4] | -2.3 [-2.3 to -2.3]
  V6: number analyzed (Participants) | 2 | 0
  V6 | -1.45 [-1.9 to -1] |

10. Secondary Outcome: Warmth Detection Threshold (WDT)
Description: Change of Warmth Detection Threshold from V1 to V6 The Warmth Detection Threshold (WDT) was measured according to the established protocol of Deutscher Forschungsverbund Neuropathischer Schmerz (DFNS). See Rolke, R et al. "Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values." Pain vol. 123,3 (2006): 231.
  Raw data were z-transformed by subtracting the mean value of the corresponding reference group followed by a division the respective standard deviation. If the resulting z-value exceeds 1.96, it is outside the 95% confidence interval of the standard normal distribution with zero mean and unit variance, independent of the original units of measurement.
  (also see Rolke et. al.). A higher z-value indicates an improvement.
Time Frame: day 0 (baseline) and day 78 (V6; 10 weeks)
Population: Due to low number of participants only descriptive data is available
Measure: Mean (Full Range); unit: Z-score
Arm/Group | Oxycodone | Tapentadol
Number analyzed (Participants) | 1 | 2
Z-score
  V1 | -2 [-2 to -2] | -1.05 [-2 to -0.1]
  V6: number analyzed (Participants) | 0 | 2
  V6 |  | -2 [-2.2 to -1.8]

11. Secondary Outcome: Thermal Sensory Limen (TSL)
Description: Change of Thermal Sensory Limen from V1 to V6 The Thermal Sensory Limen (TSL) was measured according to the established protocol of Deutscher Forschungsverbund Neuropathischer Schmerz (DFNS). See Rolke, R et al. "Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values." Pain vol. 123,3 (2006): 231.
  Logarithmically trasnformed raw data were z-transformed by subtracting the mean value of the corresponding reference group followed by a division the respective standard deviation. If the resulting z-value exceeds 1.96, it is outside the 95% confidence interval of the standard normal distribution with zero mean and unit variance, independent of the original units of measurement.
  (also see Rolke et. al.). A higher z-value indicates an improvement.
Time Frame: day 0 (baseline) and day 78 (V6; 10 weeks)
Population: Due to low number of participants only descriptive data is available
Measure: Mean (Full Range); unit: Z-score
Arm/Group | Oxycodone | Tapentadol
Number analyzed (Participants) | 1 | 2
Z-score
  V1 | -2.1 [-2.1 to -2.1] | -1.9 [-3.9 to 0.1]
  V6: number analyzed (Participants) | 0 | 2
  V6 |  | -2.45 [-2.6 to -2.3]

12. Secondary Outcome: Mechanical Detection Threshold (MDT)
Description: Change of Mechanical Detection Threshold from V1 to V6 The Mechanical Detection Threshold (MDT) was measured according to the established protocol of Deutscher Forschungsverbund Neuropathischer Schmerz (DFNS). See Rolke, R et al. "Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values." Pain vol. 123,3 (2006): 231.
  Logarithmically transformed raw data were z-transformed by subtracting the mean value of the corresponding reference group followed by a division the respective standard deviation. If the resulting z-value exceeds 1.96, it is outside the 95% confidence interval of the standard normal distribution with zero mean and unit variance, independent of the original units of measurement.
  (also see Rolke et. al.). A higher z-value indicates an improvement.
Time Frame: day 0 (baseline) and day 78 (V6; 10 weeks)
Population: Due to low number of participants only descriptive data is available
Measure: Mean (Full Range); unit: Z-score
Arm/Group | Oxycodone | Tapentadol
Number analyzed (Participants) | 1 | 2
Z-score
  V1 | -2.2 [-2.2 to -2.2] | -0.1 [-0.2 to 0]
  V6: number analyzed (Participants) | 0 | 2
  V6 |  | -1 [-2.1 to 1]

13. Secondary Outcome: Vibration Detection Threshold (VDT)
Description: Change of Vibration Detection Threshold from V1 to V6 The Vibration Detection Threshold (VDT) was measured according to the established protocol of Deutscher Forschungsverbund Neuropathischer Schmerz (DFNS). See Rolke, R et al. "Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values." Pain vol. 123,3 (2006): 231.
  Raw data were z-transformed by subtracting the mean value of the corresponding reference group followed by a division the respective standard deviation. If the resulting z-value exceeds 1.96, it is outside the 95% confidence interval of the standard normal distribution with zero mean and unit variance, independent of the original units of measurement.
  (also see Rolke et. al.). A higher z-value indicates an improvement.
Time Frame: day 0 (baseline) and day 78 (V6; 10 weeks)
Population: Due to low number of participants only descriptive data is available
Measure: Mean (Full Range); unit: Z-score
Arm/Group | Oxycodone | Tapentadol
Number analyzed (Participants) | 1 | 2
Z-score
  V1 | -1.8 [-1.8 to -1.8] | -1.85 [-4.8 to -1.1]
  V6: number analyzed (Participants) | 0 | 2
  V6 |  | -1.72 [-3.3 to 0]

14. Secondary Outcome: Paradoxical Heat Sensations (PHS)
Description: Change of Number of Paradoxical Heat Sensations from V1 to V6 The number of Paradoxical Heat Sensations (PHS) was measured according to the established protocol of Deutscher Forschungsverbund Neuropathischer Schmerz (DFNS). See Rolke, R et al. "Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values." Pain vol. 123,3 (2006): 231.
  An occurence of up to three paradoxical heat sensations was possible. The number was assessed. A lower number indicates an improvement.
Time Frame: day 0 (baseline) and day 78 (V6; 10 weeks)
Population: Due to low number of participants only descriptive data is available
Measure: Mean (Full Range); unit: sensations out of 3
Arm/Group | Oxycodone | Tapentadol
Number analyzed (Participants) | 1 | 2
sensations out of 3
  V1 | 0 [0 to 0] | 0.5 [0 to 1]
  V6: number analyzed (Participants) | 0 | 2
  V6 |  | 0 [0 to 0]

ADVERSE EVENTS:
Groups:
- Tapentadol Retard: daily dose of max. 500 mg and min. 200 mg
- Oxycodon Retard: daily dose of max. 120 mg and min. 40 mg
Arm/Group | Tapentadol Retard | Oxycodon Retard
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tapentadol Retard (N=2) | Oxycodon Retard (N=1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting/nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
fatigue (General disorders) | 1 | 0
pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
swollen, red, hot left knee (Musculoskeletal and connective tissue disorders) | 1 | 0
dizzieness (Nervous system disorders) | 0 | 1
hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
difficulty concentrating (Nervous system disorders) | 0 | 1
eczema of the left hand (Skin and subcutaneous tissue disorders) | 1 | 0
headache (Nervous system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes